CLINICAL TRIAL: NCT05774639
Title: A Randomized, Multicenter, Double-Blind, 4-Arm, Parallel-Group, Active Controlled, Phase 3 Study to Compare Efficacy, Safety and Immunogenicity of ADL-018 150 mg and 300 mg With US-Licensed Xolair® 150 mg and 300 mg Administered Through Subcutaneous Route Every 4 Weeks in Patients With Chronic Idiopathic Urticaria (CIU) Who Remained Symptomatic Despite Treatment With Approved Doses of H1 Antihistamines
Brief Title: Study to Compare Efficacy Safety and Immunogenicity of ADL-018 With XOLAIR (Omalizumab) in Adults With Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Collaborators: COD Research Private Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBS/OMA/01
Record Dates: First submitted 2023-02-25; First posted 2023-03-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: This will be parallel study to compare efficacy, safety and immunogenicity of ADL-018 150 and 300 mg doses in comparison with US-licensed XOLAIR 150 and 300 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- ADL-018 300 mg Main Treatment period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 0, 4, 8
  Interventions: Drug: Omalizumab Injection
- Xolair-300 mg Main Treatment Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 0, 4, 8
  Interventions: Drug: Xolair Prefilled Syringe
- ADL-018 150 mg Main Treatment period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 0, 4, 8
  Interventions: Drug: Omalizumab Injection
- Xolair-150 mg Main Treatment Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 0, 4, 8
  Interventions: Drug: Xolair Prefilled Syringe
- ADL-018 300 mg Main / ADL-018 300 mg Transition Period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to ADL-018 300 mg in the Main Treatment period.
  Interventions: Drug: Omalizumab Injection
- Xolair-300 mg Main / ADL-018 300 mg Transition Period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to Xolair-300 mg in the main treatment period.
  Interventions: Drug: Omalizumab Injection; Drug: Xolair Prefilled Syringe
- Xolair-300 mg Main / Xolair-300 mg Transition Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered twice (total dosage 300 mg) at week 12,16,20 in patients that were randomized to Xolair-300 mg in the main treatment period.
  Interventions: Drug: Xolair Prefilled Syringe
- ADL-018 150 mg Main / ADL-018 150 mg Transition Period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to ADL-018150 mg in the main treatment period.
  Interventions: Drug: Omalizumab Injection
- Xolair-150 mg Main / ADL-018150 mg Transition Period (Experimental): ADL-018 (Omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to XOLAIR-150 mg in the main treatment period.
  Interventions: Drug: Omalizumab Injection; Drug: Xolair Prefilled Syringe
- Xolair-150 mg Main / Xolair-150 mg Transition Period (Active Comparator): XOLAIR (omalizumab) injection 150 mg/mL pre-filled syringe administered with one placebo injection at week 12,16,20 in patients that were randomized to XOLAIR -150 mg in the main treatment period.
  Interventions: Drug: Xolair Prefilled Syringe

INTERVENTIONS:
Drug: Omalizumab Injection — ADL-018 (Omalizumab) solution for injection 150 mg/mL prefilled syringe (PFS)
  Other Names: ADL-018
  Arms: ADL-018 150 mg Main / ADL-018 150 mg Transition Period; ADL-018 150 mg Main Treatment period; ADL-018 300 mg Main / ADL-018 300 mg Transition Period; ADL-018 300 mg Main Treatment period; Xolair-150 mg Main / ADL-018150 mg Transition Period; Xolair-300 mg Main / ADL-018 300 mg Transition Period
Drug: Xolair Prefilled Syringe — XOLAIR (omalizumab) injection is supplied as a single dose PFS. Each PFS of XOLAIR contains 150 mg of omalizumab in 1 mL of solution
  Arms: Xolair-150 mg Main / ADL-018150 mg Transition Period; Xolair-150 mg Main / Xolair-150 mg Transition Period; Xolair-150 mg Main Treatment Period; Xolair-300 mg Main / ADL-018 300 mg Transition Period; Xolair-300 mg Main / Xolair-300 mg Transition Period; Xolair-300 mg Main Treatment Period

SUMMARY:
The purpose of the study is to compare the efficacy, safety, tolerability, and immunogenicity of ADL-018 compared to XOLAIR in patients with Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) who remain symptomatic on H1 antihistamine treatment

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind study to demonstrate similar efficacy and safety of ADL-018 compared to XOLAIR administered sc at doses of 300 mg or 150 mg every 4 weeks for 24 weeks (6 treatments) in patients with Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) who remain symptomatic despite antihistamine (H1) treatment. This study will consist of a screening period (up to 2 weeks), a 24-week treatment period consisting of a 12-week double-blind main treatment period and a 12-week double-blind transition period, which is followed by a 16-week follow-up period. The total duration of the study is up to 42 weeks.

At baseline, patients will be randomized in a 2:2:1:1 ratio to receive the first 3 treatments of ADL-018 300 mg, XOLAIR 300 mg, ADL-018 150 mg or XOLAIR 150 mg (main treatment period). At Week 12, prior to receiving their fourth dose of study medication, patients in the XOLAIR 300 mg and the XOLAIR 150 mg treatment groups will be randomized 1:1 to receive 3 additional doses of XOLAIR (at the same dose level as prior to randomization, or switch to 3 doses of ADL-018 (transition period) at the same dose level as prior to randomization. All patients in the ADL-018 groups will continue to receive ADL-018 at the same dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written informed consent, adhering to all visit schedules, and meeting study requirements.
2. Male or female patients 18 to 75 years of age (both inclusive) at the time of screening.
3. Diagnosis of CIU refractory to H1 antihistamines at the time of randomization, as defined by all of the following:

   * CIU diagnosis for at least 6 months.
   * Must have been on an approved H1 antihistamine for CIU for at least 3 consecutive days immediately prior to the Day -14 screening visit and must document current use on the day of initial screening.
   * Presence of itch and hives for ≥ 8 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamine treatment.
   * In-clinic UAS ≥ 4 on at least 1 of the screening visit days (Day -14, Day -7, or Day 1).
   * UAS7 (range 0-42) ≥ 16 and itch component of UAS7 (range 0-21) ≥ 8 during 7 days prior to randomization.
4. Willing and able to complete a daily symptom diary for the duration of the study and must not have any missing diary entries in the 7 days prior to randomization.
5. Females of childbearing potential must be willing to use acceptable contraceptive methods throughout the study and for 6 months thereafter.
6. Females of non-childbearing potential must have undergone sterilization procedures, at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone serum levels consistent with postmenopausal status.

Exclusion Criteria:

1. Participation in a clinical trial involving the administration of an investigational drug or marketed drug within 30 days prior to initial dosing (90 days for biologics).
2. Clearly defined underlying etiology for chronic urticarias other than CIU.
3. Evidence of parasitic infection.
4. Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or any other skin disease associated with itch.
5. Previous treatment with omalizumab within a year prior to screening.
6. Routine doses of the following medications within 10 days prior to screening: Systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide or investigational agents such as benralizumab or dupilumab etc.
7. IVIG ( Intravenous immune globulin) or plasmapheresis within 90 days prior to screening.
8. Regular (daily/every other day) doxepin (oral) use within 14 days prior to screening.
9. Any H2 antihistamine use within 7 days prior to screening.
10. Any LTRA (Leukotriene receptor antagonists such as montelukast or zafirlukast) within 10 to 14 days prior to screening.
11. Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.
12. Hypersensitivity to omalizumab or any component of the formulation.
13. History of anaphylactic shock.
14. Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic, or other pathological conditions that could interfere with the interpretation of the study results and/or compromise the safety of the patients.
15. Medical examination or laboratory findings that suggest the possibility of decompensation of co-existing conditions for the duration of the study.
16. Evidence of current drug or alcohol abuse.
17. Positive test for hepatitis B, hepatitis C, or HIV.
18. Females with positive pregnancy tests at screening or any other visit.
19. Females who are breastfeeding or lactating.
20. History of any clinically significant disease or condition that, in the opinion of the Principal Investigator (PI)/designee, would render them unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the ISS7 at Week 12 between ADL-018 300 mg and XOLAIR 300 mg | Change from Baseline at week 12
  ISS 7 is a weekly itch severity score calculated as sum of the daily itch severity score for 7 days, on a scale of 0 to 3 (0=none to 3=intense/severe)
Relative potency of ADL-018 and XOLAIR | Change from Baseline at week 12
  Relative potency ADL-018 to the Xolair defined as the dose of ADL-018 that produces the same biological response as one unit of the dose of the Xolair.
  The relative potency and its CI will be measured by change in ISS7 at Week 12 using a 4 point assay based on the 300 mg and 150 mg dose levels of each product.

SECONDARY OUTCOMES:
Change from baseline in the ISS7 at Week 2, 4, 6, 8, 16, 20, and 24 | Change from Baseline at Week 2, 4, 6, 8, 16, 20, and 24
  ISS 7 is a weekly itch severity score calculated as sum of the daily itch severity score for 7 days, on a scale of 0 to 3 (0=none to 3=intense/severe).
Change from baseline in UAS7 at Weeks 2, 4, 6, 8, 12, 16, 20, and 24 | Change from Baseline at Weeks 2, 4, 6, 8, 12, 16, 20, and 24
  Change from baseline in the Urticaria Activity Score (UAS) - sum of the daily number of wheals score and itch severity score over 7 days, range from 0 (minimum) to 6 (maximum)
Change from baseline in weekly number of hives (urticaria) score (HSS7) at Weeks 2, 4, 6, 8, 12, 16, 20, and 24 | Change from Baseline at Weeks 2, 4, 6, 8, 12, 16, 20, and 24.
  Change from baseline in the weekly number of wheals score at Week 12
Percentage of patients with angioedema-free days from Week 4 to Week 12 | change from Week 4 to Week 12
  Percentage of angioedema-free days from Week 4 to Week 12
Percentage of complete responders (UAS7=0) at Week 12 | change from baseline at week 12
  Percentage of complete responders with weekly Urticaria Activity Score =0 at Week 12
Percentage of patients achieving UAS7 ≤ 6 at Weeks 2, 4, 6, 8, 12, 16, 20, and 24 | Change from Baseline at Weeks 2, 4, 6, 8, 12, 16, 20, and 24
  Percentage of patients with a weekly Urticaria Activity Score ≤6
Change from baseline in the overall Dermatology Life Quality Index (DLQI) score at weeks 4, 8, 12, 16, 20, and 24. | Change from Baseline at Week 12
  Change from baseline in the overall dermatology life quality index (DLQI) score at Week 12; comparisons of ADL-018 and XOLAIR treatment arms. The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - True Blue Clinical Research, Brandon, Florida
  - Access Research Institute, Brooksville, Florida
  - San Marcus research Clinic, Inc, Miami Lakes, Florida
  - Options Research Group, West Lafayette, Indiana
- Site 001, Mumbai, Maharashtra, India
- Al Essra Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No